CLINICAL TRIAL: NCT00287183
Title: Double-Blind, Randomized, Placebo-Controlled, Phase IIa, Multicenter Study In Patients With Type 2 Diabetes And Persistent Albuminuria To Evaluate The Safety And Efficacy Of A Six Month Regimen Of Orally-Administered TTP488
Brief Title: 6-Month Safety And Efficacy Study Of TTP488 In Patients With Type 2 Diabetes And Persistent Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0341001; TTP488-202
Record Dates: First submitted 2006-01-20; First posted 2006-02-06 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — azeliragon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04494700 (TTP488) (Active Comparator)
  Interventions: Drug: PF-04494700 (TTP488)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-04494700 (TTP488) — 60 mg/day for 6 days followed by 20 mg/day for 175 days vs placebo, oral medication
  Arms: PF-04494700 (TTP488)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Current research indicates that TTP488 may be a viable agent for the treatment of diabetic nephropathy. The purpose of this study is to determine the safety and efficacy of a six-month regimen of daily orally-administered TTP488 to patients with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 31 years of age or older.
* Females must no longer be of child-bearing potential, must have a negative serum pregnancy test, and cannot be breast-feeding.
* Non-vasectomized male must be willing to abstain from sexual intercourse or willing to use a condom in addition to having their female partner use another form of contraception.
* Diagnosis of probable Type 2 diabetes after the age of 30 and for at least 6 months prior to the screening visit and: not requiring insulin within first year of diagnosis; no history of diabetic ketoacidosis (DKA); body mass index (BMI) of 40 or less at the screening visit
* Presence of persistent albuminuria with a UACR of 6.7 - 203 mg/mmol Must be taking the highest tolerated dose of an angiotensin converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB) and have been maintained on that dose for at least 3 months prior to the Baseline visit
* Blood pressure(BP) must be stable and well controlled by the judgement of the investigator (goal of the control of BP is 130/80 or less). If required, the use of anti-hypertensives in addition to an ACE inhibitor or an ARB is acceptable.
* Patients with a calculated creatinine clearance of greater than or equal to 30 mL/min and without the presence of clinically significant hematuria or red or white cell casts can be included in the study.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes
* Hemoglobin A1c (HbA1c) >10%
* Females cannot be breast-feeding
* Known renal artery stenosis
* Calculated creatinine clearance <30 mL/min or the presence of clinically significant hematuria of red or white cell casts
* Chronic use of NSAIDs or more than 1 g/day of aspirin
* QTc >450 msec for females or >430 msec for males (a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle)
* Known family history of prolonged QT syndrome
* History of symptomatic congestive heart failure within the last 2 years
* History of syncope in the lst 2 years or recurrent hypokalemia, including that caused by diuretics
* Myocardial infarction or signs or symptoms of unstable coronary artery disease with the last year
* Pulmonary disease or evidence of clinically significant pulmonary symptoms.
* Active neoplastic disease. (Excised cutaneous basal cell carcinomas are not excluded). Patients with stable prostate cancer may be included at the discretion of the Medical Monitor.
* Any clinically significant hematologic or coagulation disorder
* Any clinically significant hepatic disease
* Use of excluded medications: drugs known to significantly increase QTc and/or have increased risk of torsades de point, immunosuppressive agents, cancer chemotherapeutic agents, oral corticosteroids other than maintenance doses equivalent to 7.5 mg prednisone per day, and radiotherapy
* Use of an investigational drug within 30 days or within 5 half-lives of the investigational agent, whichever is longer, or use of an investigational medical device within 2 weeks before or after the study
* Any other disease or condition that, in the opinion of the investigator, makes the patient unsuitable to participate in this study

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary endpoint of efficacy will be assessed by comparing the treatment groups based on the change in urinary albumin-creatinine ratio (UACR) | from baseline to end of treatment (Month 6).

SECONDARY OUTCOMES:
To evaluate treatment on estimated GFR and serum creatinine | evaluated for change from baseline to months 3 & 6
To evaluate the effects of TTP488 on other relevant biomarkers | evaluated at months 1, 3 & 6
To evaluate the safety of TTP488 | Ongoing
To evaluate the PK profile of oral TTP488. | Ongoing
To evaluate the effect of treatment with TTP488 on UACR | evaluated from baseline to month 3 visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Canada (17):
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Penticton, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Courtice, Ontario
  - Pfizer Investigational Site, Fort Erie, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Millon, Ontario
  - Pfizer Investigational Site, North Bay, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Saint Catherines, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Smith Falls, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0341001&StudyName=6-Month%20Safety%20And%20Efficacy%20Study%20Of%20TTP488%20In%20Patients%20With%20Type%202%20Diabetes%20And%20Persistent%20Albuminuria